CLINICAL TRIAL: NCT01271582
Title: Investigation of Association Between UGT1A1 Polymorphisms and Irinotecan Toxicity in Korean Patients With Advanced Colorectal or Gastric Cancer Treated With FOLFIRI Regimen
Brief Title: Investigation of Association Between UGT1A1 Polymorphisms and Irinotecan Toxicity in Korean Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Tae Won Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPT_08_001
Record Dates: First submitted 2011-01-04; First posted 2011-01-07 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Stage IV Colorectal Cancer; Gastric Cancer
Keywords: Colorecatal cancer; Gastric cancer; Irinotecan; UGT1A1; Neutropenia
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Neutropenia | interventions — Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFIRI (Experimental): Patients with colorectal cancer or gastric cancer will be treated with FOLFIRI(Irinotecan, 5FU, leucovorin) regimen upto 12 cycles. (Single arm study)
  Interventions: Drug: Irinotecan, 5FU, leucovorin

INTERVENTIONS:
Drug: Irinotecan, 5FU, leucovorin — FOLFIRI regimen every 2 weeks [irinotecan 150mg/m2 or 180mg/m2, leucovorin 20(200)mg/m2, 5FU 400 mg/m2 (bolus) or 2400 mg/m2 (46hour infusion)]
  Other Names: CAMPTO (CAMPOSAR)

SUMMARY:
The purpose of this study is to investigate the association between UGT1A1 polymorphisms and neutropenia and diarrhea in Korean patients with advanced colorectal or gastric cancer treated with FOLFIRI regimen.

ELIGIBILITY:
Inclusion Criteria:Subjects should meet all of the following criteria to participate in the trial.

* Histologically confirmed colorectal or gastric cancer patients who are chemonaive or failed to 1st line chemotherapy
* Subjects who are expected to receive toxicity test at least once after FOLFIRI treatment.
* Aged 18 years or older.
* ECOG performance status of ≤ 2.
* Anticipated life expectancy of ≥ 3 months.
* Clinically acceptable function of bone marrow, kidney and liver function as below.

  1. ANC ≥ 1500/mm3 and platelet count ≥ 100,000/mm3
  2. Serum total bilirubin ≤ 1.5 x ULN, alkaline phosphatase ≤ 2.5 x ULN, Serum ALT and AST ≤ 2.5 x ULN (Serum ALT and AST ≤ 5 x ULN, if liver metastases are present)
  3. Serum creatinine ≤ 1.5 mg/dL or CLcr > 60 ml/min
* Subjects whose written informed consent can be obtained prior to their participation in the trial.

Exclusion Criteria: Subjects who meet any of the following criteria should not be included in the trial.

* Pregnant or breast feeding women
* Serious concurrent complication, severe active infection.
* Subjects with chronic diarrhea, paralytic ileums, pulmonary fibrosis or pneumonia interstitialis
* Subjects with epilepsia or severe psychiatric disorders.
* Subjects who are regarded to be unsuitable for this trial by the investigator.
* Subjects who are participating in other clinical trials
* Subjects who have received prior chemotherapy including irinotecan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-06 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Association between UGT1A1 polymorphism and grade 3/4 neutropenia after 1st cycle of FOLFIRI treatment | 2 weeks
  During the first cycle of treatment

SECONDARY OUTCOMES:
Association between UGT1A1 polymorphism and grade 3/4 neutropenia in all treatment duration | 24 weeks
  During all treatment period(during 12 cycle, each 2 weeks)
Association between grade 3/4 diarrhea and UGT1A1 polymorphism | 2 weeks
  During the first cycle of treatment
Progression-free survival | 6 months (average)
  The time from registration to objective tumor progression or death

CONTACTS AND LOCATIONS:
Overall Officials: YongSang Hong, Professor, Study Director — Asan Medical Center
Locations (5):
- South Korea (5):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Hwasun Hospital, Jeonam, Hwasun-gun
  - Korea Cancer Center Hospital, Seoul, Nowon-Gu
  - Asan Medical Center, Seoul, Songpa-Gu
  - National Cancer Center, Goyang